CLINICAL TRIAL: NCT00482976
Title: The Effects of a Protein Kinase C Beta Inhibitor, LY333531, on Vascular and Neural Functions in Type 2 Diabetes Mellitus - Study B7A-MC-MBDM
Brief Title: Effect of LY333531 on Vascular and Neural Functions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chromaderm, Inc. (Industry)
Collaborators: Joslin Diabetes Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 7546; B7A-MC-MBDM
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — ruboxistaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ruboxistaurin
Drug: Placebo

SUMMARY:
To determine if protein kinase C beta plays a significant role in vascular endothelial dysfunction, small fiber neural dysfunction, and oxidative stress associated with diabetes mellitus.

DETAILED DESCRIPTION:
32mg Ruboxistaurin; 4 week cross-over treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed for at least 1 mo and less than 10 yrs prior to visit 1
* HbA1c less than 9% and fasting plasma glucose less than 260mg/dl
* Blood pressure less than 160/100 mmHg
* Total cholesterol less than 300 mg/dl and/or triglycerides less than 600 mg/dl

Exclusion Criteria:

* Subjects treated with a thiazolidinedione (TZD) in 12 weeks prior to visit 1.
* History of heart disease (MI, unstable angina, CVA, TIA, CABG, or percutaneous transluminal coronary angioplasty) w/in 6 months of visit 1 or subjects with BYHA class III or IV congestive heart failure.
* Female subjects of child-bearing potential that are pregnant or intend to become pregnant (i.e. not practicing an acceptable method of birth control)
* TSH greater than 1.5 times upper limit of normal at V1 or other endocrine disease.
* ALT greater than 1.5 times upper limit of normal at V1; Serum creatinine greater than 2.0mg/dl at V1; micro-albumin greater than 300.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-12; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Improvement in endothelium-dependent vasodilation of the microcirculation of the skin and nerve axon-related reflex vasodilation. | 4 weeks
Improvement in endothelium-dependent vasodilation of the brachial artery (flow mediated dilation) | 4 weeks
Improvement in selective measurements of oxidative stress, endothelial activity and vascular abnormalities which will correlate with PKC activity in the peripheral monocytes. | 4 weeks

SECONDARY OUTCOMES:
Safety of ruboxistaurin | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com